CLINICAL TRIAL: NCT01147952
Title: A Randomised Trial of the Effect of Exercise on Peripheral Blood Gene Expression in Patients With Stable Angina
Brief Title: The Effect of Exercise on Peripheral Blood Gene Expression in Angina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STH15565
Record Dates: First submitted 2010-06-18; First posted 2010-06-22 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Angina Pectoris
Keywords: angina; gene expression; depression; anxiety
MeSH Terms: conditions — Angina Pectoris; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 12 week exercise training (Experimental)
  Interventions: Behavioral: Structured exercise training
- Conventional Care (No Intervention)

INTERVENTIONS:
Behavioral: Structured exercise training — randomised to 12 weeks of exercise training up to three times weekly. Training will be interval training with active recovery, with 3 min intervals conducted 10bpm below angina threshold.
  Arms: 12 week exercise training

SUMMARY:
Regular exercise is known to produce significant health benefits and to reduce the risk of heart diseases, although how this benefit occurs is not well understood. White blood cells are known to be involved in triggering heart attacks, and which genes are switched on or off in white blood cells determines whether they have beneficial or harmful effects. Previous studies, and studies ongoing in our group, have demonstrated measurement of peripheral blood gene expression (which reflects white blood cell gene expression) is able to distinguish between patients with and without coronary artery disease, or patients who are able to develop good compared with poor coronary collateral arteries. Therefore, the gene expression signature in peripheral blood may provide novel diagnostic or prognostic information, and insight into the pathogenesis of heart disease.

We therefore hypothesise that exercise alters peripheral blood gene expression in patients with coronary artery disease and angina. This will identify possible ways that exercise improves angina and reduces the risk of heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Class I to III angina pectoris (classified according to the Canadian Cardiovascular Society [CCS])with documented myocardial ischemia or coronary artery disease on angiography
* Ability to read and speak English to a level allowing satisfactory completion of written questionnaires and to understand instruction during the exercise programme.

Exclusion Criteria:

* Acute coronary syndromes or recent myocardial infarction (<2 months)
* Left main coronary artery stenosis >25% or high-grade proximal left anterior descending artery stenosis
* Known reduced left ventricular function (ejection fraction <40%)
* Significant valvular heart disease
* Insulin-dependent diabetes mellitus
* Occupational, orthopedic, and other conditions that preclude regular exercise
* Patients whose ECG prevents interpretation of an exercise test (LBBB, RBBB, pacemaker implantation).
* Patients who already perform greater than 30min continuous exercise three times weekly (self-reported).

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Peripheral blood gene expression | baseline
Peripheral blood gene expression | 6wks after starting 12week exercise training (or conventional care)
peripheral blood gene expression | 12 weeks after exercise training (or conventional care)
Peripheral blood gene expression | 24 weeks after starting 12 weeks exercise training programme

SECONDARY OUTCOMES:
Angina status | baseline
Angina status | 6wks after starting 12 week exercise programme (or conventional care)
Angina status | 12wks after starting 12 week exercise programme (or conventional care)
Angina Status | 24wks after starting 12 week exercise programme (or conventional care)
Anxiety Score | baseline
Anxiety Score | 6wks after starting 12 week exercise programme (or conventional care)
Anxiety Score | 12wks after starting 12 week exercise programme (or conventional care)
Anxiety Score | 24wks after starting 12 week exercise programme (or conventional care)
Depression Score | 6wks after starting 12 week exercise programme (or conventional care)
Depression Score | baseline
Depression Score | 12wks after starting 12 week exercise programme (or conventional care)
Depression Score | 24wks after starting 12 week exercise programme (or conventional care)

CONTACTS AND LOCATIONS:
Locations (1):
- NIHR Cardiovascular Biomedical Research Unit, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bourke L, Tew GA, Milo M, Crossman DC, Saxton JM, Chico TJ. Study protocol: a randomised controlled trial investigating the effect of exercise training on peripheral blood gene expression in patients with stable angina. BMC Public Health. 2010 Oct 18;10:620. doi: 10.1186/1471-2458-10-620. PMID 20955605